CLINICAL TRIAL: NCT02093169
Title: Interventional, Open-label, Positron Emission Tomography (PET) Study Investigating D2 Dopamine Receptor Occupancy After Oral Dosing of Lu AF35700 in Healthy Men Using [11C]-PHNO as Tracer Compound
Brief Title: D2 Dopamine Receptor Occupancy After Oral Dosing of Lu AF35700 in Healthy Men Using [11C]-PHNO as Tracer Compound
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15868A; 2013-004283-61 (EudraCT Number)
Record Dates: First submitted 2014-03-19; First posted 2014-03-20 (Estimated); Last update posted 2014-09-23 (Estimated); Status verified 2014-09

CONDITIONS: Healthy Men

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part A: Lu AF35700 (Experimental)
  Interventions: Drug: Part A: Lu AF35700
- Part B: Lu AF35700 (Experimental)
  Interventions: Drug: Part B: Lu AF35700

INTERVENTIONS:
Drug: Part A: Lu AF35700 — One 30 mg single dose for one day; orally
  Arms: Part A: Lu AF35700
Drug: Part B: Lu AF35700 — Daily dosing: 10 mg for 3 days, 20 mg for 3 days, 45 mg on Day 7; orally
  Arms: Part B: Lu AF35700

SUMMARY:
To investigate the relationship between the combined Lu AF35700 and Lu AF36152 plasma concentration and D2 dopamine receptor occupancy up to 172 hours after oral dosing of Lu AF35700

ELIGIBILITY:
Inclusion Criteria:

* Healthy young men >=25 and <=45 years of age with a Body Mass Index (BMI) >=18.5 kg/m2 and <=30 kg/m2.

Other protocol-defined Inclusion and Exclusion criteria may apply.

Ages: 25 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-02; Primary Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Relationship between plasma concentrations and pharmacodynamic (PD) measures specified as binding potential at each scanning time point | Up to 172 hours after dosing
Relationship between plasma concentrations and PD measures specified as plasma concentrations of Lu AF35700, Lu AF36152 and Lu AF35700 + Lu AF36152 at each scanning time point | Up to 172 hours after dosing
Relationship between plasma concentrations and PD measures specified as occupancy in relation to plasma concentrations of Lu AF35700, Lu AF36152 and Lu AF35700 + Lu AF36152, respectively | Up to 172 hours after dosing

SECONDARY OUTCOMES:
Adverse events | Up to Week 12
Columbia Suicide Severity Rating Scale (C-SSRS) (Part B only) | Up to Week 12
Area under the curve (AUC), maximum observed concentration (Cmax), oral clearance (CL/F), and apparent elimination half-life (t½) | Up to 168 hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (1):
- GB801, London, United Kingdom